CLINICAL TRIAL: NCT01001286
Title: Questscope Non-Formal Education Impact Study
Acronym: QSNFEIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Matthew Morton, Researcher, University of Oxford, Centre for Evidence-Based Intervention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QS-001
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Education; Empowerment; Self-efficacy
Keywords: dropout youth in low income communities in Amman, Jordan
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Youth Club (Active Comparator): The intervention will be compared to a waitlist comparison group. The group will enter NFE after the four-month posttest. During the four months, the youth will be offered a biweekly recreational youth club. The club will be led by Jordanian university student volunteers out of community-based organizations. Club activities will take place approximately every two weeks, including games, sports, arts and crafts, cultural activities, and trips. The Club will not include any significant education components or youth empowerment methodology--the hypothesized active ingredients of QS NFE.
  Interventions: Behavioral: Questscope Non-Formal Education
- Questscope Non-Formal Education (Experimental): Participation in two-hour classes for three to five days per week. Duration involves 24 months of programming (three, eight-month learning cycles), but this randomized controlled trial will only assess impacts of participation in the first four months.
  Regular presence of trained, supportive adults. Educational topics and class activities determined by the youth as a group with the support of the adult teachers ("facilitators").
  Interventions: Behavioral: Questscope Non-Formal Education

INTERVENTIONS:
Behavioral: Questscope Non-Formal Education — Participation in two-hour classes for three to five days per week. Duration involves 24 months of programming (three, eight-month learning cycles), but this randomized controlled trial will only assess impacts of participation in the first four months.
  Regular presence of trained, supportive adults. Educational topics and class activities determined by the youth as a group with the support of the adult teachers ("facilitators").

SUMMARY:
This randomized controlled trial (RCT) evaluates the effectiveness of Questscope Non-Formal Education (QS NFE) on impacting psychosocial outcomes for out-of-school youth, ages 13-21, in Jordan. QS NFE is an empowerment-based education program. A unique agreement with the Jordanian Ministry of Education enables participating youth to receive a 10th-grade equivalent certificate upon successful completion of the 24-month non-formal education. The main components of QS NFE include retraining formal education teachers for fostering positive relationships with at-risk youth, asset-building learning and social activities, and a youth-driven learning environment.

The study hypothesis is that by engaging youth in positive relationships with local teachers and enabling the youth to drive the learning experience, the intervention will have positive impacts on general self-efficacy, social supports, social skills, and strengths and difficulties.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) evaluates the effectiveness of Questscope Non-Formal Education (QS NFE) on impacting psychosocial outcomes for out-of-school youth, ages 13-21, in Jordan. QS NFE is an empowerment-based education program. A unique agreement with the Jordanian Ministry of Education enables participating youth to receive a 10th-grade equivalent certificate upon successful completion of the 24-month non-formal education. The main components of QS NFE include retraining formal education teachers for fostering positive relationships with at-risk youth, asset-building learning and social activities, and a youth-driven learning environment.

The study hypothesis is that by engaging youth in positive relationships with local teachers and enabling the youth to drive the learning experience, the intervention will have positive impacts on general self-efficacy, social supports, social skills, and strengths and difficulties.

Youth will be recruited according to normal Questscope recruitment procedures by program leaders in five poverty pocket communities in Amman, Jordan. Six QS NFE centers will be involved in the impact evaluation (four male centers and 2 female centers). Youth will be recruited, enrolled, and randomized on an individual basis until each NFE center's sample target is met (between 24 and 40 youth, depending on the center). The overall sample target is 200 for the six NFE centers aggregately (100 intervention group and 100 waitlist comparison). The study aims to recruit 54 females and 146 males.

Randomization will be conducted electronically using a random permuted block method through SealedEnvelope.com. Data collection for outcome measures will involve a computer-based, self-administered questionnaire designed with The Survey System software by Creative Research Systems. The computer-based survey will provide both text and audio to accommodate low literacy levels.

In the event that a participant rejects his/her random assignment within 48 hours of enrollment, the youth will be replaced in the study and will not be included in final data analysis. Additionally, all siblings recruited together into the study will be blocked and randomized together in enrollment.

ELIGIBILITY:
Inclusion Criteria:

* age 13-18 males or 13-21 females
* out of the formal education system for more than six months

Exclusion Criteria:

* has already participated in QS NFE
* not in the above-specified age range

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
self-reported general self-efficacy | pretest at enrollment (October 2009-January 2010) and 4 months following pretest
self-reported social skills | pretest at enrollment (October 2009-January 2010) and 4 months following pretest
self-reported strengths and difficulties | pretest at enrollment (October 2009-January 2010) and 4 months following pretest
self-reported social supports | pretest at enrollment (October 2009-January 2010) and 4 months following pretest

CONTACTS AND LOCATIONS:
Locations (6):
- Jordan (6):
  - Al Mutasm School, Amman
  - Al Urdan School, Amman
  - Al Zubaidieh School, Amman
  - Ali Reda Al Rekabi School, Amman
  - Mauth Bin Jabal School, Amman
  - Umama Bint Abi Al A'as, Amman

REFERENCES:
- See also: Wesbsite for Questscope, the organization implementing the intervention. — http://www.questscope.org/